CLINICAL TRIAL: NCT07247045
Title: SuperAssist: Client-Centered Supervision Assist App for Mental Health Providers to Improve Job Well-being and Quality of Care
Brief Title: SuperAssist: Client-Centered Supervision Assist App for Mental Health Providers
Acronym: SuperAssist
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sadaaki Fukui, Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21929; R34MH133664 (NIH)
Record Dates: First submitted 2025-11-19; First posted 2025-11-25 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Behavioral Health Client-centered Supervision
Keywords: client-centered supervision, supervision, behavioral health, mobile app

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SuperAssist Group-Behavioral Health Staff (Experimental): Client-centered supervision training and use of a mobile app for behavioral health staff
  Interventions: Other: Client-centered supervision training and use of a mobile app
- Control Group-Behavioral Health Staff (No Intervention)
- SuperAssist Group-Clients (Experimental): Clients of behavioral health staff assigned to the Experimental Arm
  Interventions: Other: Client-centered supervision training and use of a mobile app
- Control Group-Clients (No Intervention): Clients of behavioral health staff assigned to the Control Arm

INTERVENTIONS:
Other: Client-centered supervision training and use of a mobile app — Behavioral health staff will learn how to implement client-centered practice and supervision with SuperAssist (Supervision Assist App). SuperAssist is designed to facilitate supervision practices around clients' identified goals and needs, which may positively impact clinician job well-being (e.g., burnout, job satisfaction), professional growth, the quality of care, and eventually client outcomes.
  Other Names: SuperAssist
  Arms: SuperAssist Group-Behavioral Health Staff; SuperAssist Group-Clients

SUMMARY:
The goal of this pilot study is to test a Supervision Assist App (SuperAssist) for implementing Client-Centered Supervision (CCS) to improve supervision practices for mental health providers (providers). During previous Aims 1 and 2, a SuperAssist beta version was designed and developed before beta testing of SuperAssist with providers and supervisors. During this pilot randomized controlled trial (Aim 3), the investigators will evaluate the feasibility, preliminary outcomes, and change mechanisms of SuperAssist.

ELIGIBILITY:
Eligibility Criteria for behavioral health staff:

* A direct service/care provider providing behavioral health services to adults in recovery from mental health or substance use conditions or a supervisor of at least one direct service/care provider for adults in a behavioral health setting of a provider or providers at a behavioral health organization
* Willing and able to attend training (approximately 8 hours), install and use the app for up to approximately 6 months, and complete the other planned study procedures

Eligibility Criteria for clients:

* At least 18 years old
* An active client (at the time of enrollment) of a participating organization
* Willing and able to receive email and/or text message communication from the study team and compete 3 online surveys over the course of the study (up to approximately 6 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Perception of Supervisory Support (PSS) Scale at 3 months | measured with staff at 3 months
  The Perception of Supervisory Support (PSS) Scale assesses perceived support from the perspective of direct service providers through measuring emotional support (e.g., feel more positively about my job), support for client goal alignment (e.g., gain greater clarity on a client's goal), and support for professional development (e.g., discuss career development), along with supervisory relationships (e.g., improve relationship with my supervisor). For supervisors, items are reframed to ask how their supervisees may perceive the level of supervisory support through their supervision. The PSS Scale uses a 6-point Likert scale ranging from 1 (Never) to 6 (Always).
Change from Baseline Perception of Supervisory Support (PSS) Scale at 6 months | measured with staff at 6 months
  The Perception of Supervisory Support (PSS) Scale assesses perceived support from the perspective of direct service providers through measuring emotional support (e.g., feel more positively about my job), support for client goal alignment (e.g., gain greater clarity on a client's goal), and support for professional development (e.g., discuss career development), along with supervisory relationships (e.g., improve relationship with my supervisor). For supervisors, items are reframed to ask how their supervisees may perceive the level of supervisory support through their supervision. The PSS Scale uses a 6-point Likert scale ranging from 1 (Never) to 6 (Always).

SECONDARY OUTCOMES:
Change from baseline Role Clarity Scale at 3 months | measured with staff at 3 months
  Role clarity will be measured by 5 items, with a 5-point response measure ranging from 1 (Not at all clear) to 5 (Perfectly clear).
Change from baseline Role Clarity Scale at 6 months | measured with staff at 6 months
  Role clarity will be measured by 5 items, with a 5-point response measure ranging from 1 (Not at all clear) to 5 (Perfectly clear).
Change from baseline Maslach Burnout Inventory (MBI) at 3 months | measured with staff at 3 months
  Burnout will be measured by the 22-item Maslach Burnout Inventory, a widely-used measure that assesses emotional exhaustion, depersonalization, and personal accomplishment using a 7 point scale ranging from 0 (Never) to 6 (Every Day)
Change from baseline Maslach Burnout Inventory (MBI) at 6 months | measured with staff at 6 months
  Burnout will be measured by the 22-item Maslach Burnout Inventory, a widely-used measure that assesses emotional exhaustion, depersonalization, and personal accomplishment using a 7 point scale ranging from 0 (Never) to 6 (Every Day)
Change from baseline Turnover Intentions-Considered Leaving at 3 months | measured with staff at 3 months
  This is the first of two questions in which staff will be asked about turnover intentions. Staff will be asked, "How often have you seriously considered leaving your job in the past six months?" using a scale ranging from 1 (Never) to 6 (Several times a week).
Change from baseline Turnover Intentions-Considered Leaving at 6 months | measured with staff at 6 months
  This is the first of two questions in which staff will be asked about turnover intentions. Staff will be asked, "How often have you seriously considered leaving your job in the past six months?" using a scale ranging from 1 (Never) to 6 (Several times a week).
Change from baseline Turnover Intentions-Likely to leave at 3 months | measured with staff at 3 months
  This is the second of two questions in which staff will be asked about turnover intentions. Staff will be asked, "How likely are you to leave your job in the next six months?" using a scale ranging from 1 (Not likely at all) to 4 (Very likely).
Change from baseline Turnover Intentions-Likely to leave at 6 months | measured with staff at 6 months
  This is the second of two questions in which staff will be asked about turnover intentions. Staff will be asked, "How likely are you to leave your job in the next six months?" using a scale ranging from 1 (Not likely at all) to 4 (Very likely).
Change from baseline Job Satisfaction at 3 months | measured with staff at 3 months
  Job satisfaction will be assessed with one item from the Job Diagnostics Survey, "Overall, I am satisfied with my job," using the scale ranging from 1 (Strongly Disagree) to 7 (Strongly Agree).
Change from baseline Job Satisfaction at 6 months | measured with staff at 6 months
  Job satisfaction will be assessed with one item from the Job Diagnostics Survey, "Overall, I am satisfied with my job," using the scale ranging from 1 (Strongly Disagree) to 7 (Strongly Agree).
Change from baseline Implementation Readiness Measure at 3 months | measured with staff at 3 months
  This scale is used to evaluate the readiness and potential success of evidence-based practice implementation using a scale ranging from 1 (Completely disagree) to 5 (Completely agree).
Change from baseline Implementation Readiness Measure at 6 months | measured with staff at 6 months
  This scale is used to evaluate the readiness and potential success of evidence-based practice implementation using a scale ranging from 1 (Completely disagree) to 5 (Completely agree).
Change from baseline Person Centered Care (PCC) Subscale at 3 months | measured with staff at 3 months
  Perceived quality of care will be measured by Person Centered Care (PCC), one of the two sub-scales of the Quality of Mental Health Care Scale (clinician version) developed to assess how mental health care providers rate the quality of care they provide (e.g., I was able to support a client's action step toward a personal goal) using a scale ranging from 0 (Never) to 5 (always).
Change from baseline Person Centered Care (PCC) Subscale at 6 months | measured with staff at 6 months
  Perceived quality of care will be measured by Person Centered Care (PCC), one of the two sub-scales of the Quality of Mental Health Care Scale (clinician version) developed to assess how mental health care providers rate the quality of care they provide (e.g., I was able to support a client's action step toward a personal goal) using a scale ranging from 0 (Never) to 5 (always).
Change from baseline System Usability Scale (SUS) at 3 months | measured with staff at 3 months
  SuperAssist Usability (experimental group only) will be measured by the System Usability Scale (SUS), which consists of 10 items with 5-point response options, ranging from 1 (Completely agree) to 5 (Completely disagree).
Change from baseline System Usability Scale (SUS) at 6 months | measured with staff at 6 months
  SuperAssist Usability (experimental group only) will be measured by the System Usability Scale (SUS), which consists of 10 items with 5-point response options, ranging from 1 (Completely agree) to 5 (Completely disagree).
Change from baseline Working Alliance Inventory (WAI) at 3 months | measured with clients at 3 months
  Perceived relatedness will be assessed with this short form of the patient version of the WAI and is 12 items (e.g., We agree on what is important for me to work on.). The item scores will be averaged and the scale is 1 (Never) to 7 (Always).
Change from baseline Working Alliance Inventory (WAI) at 6 months | measured with clients at 6 months
  Perceived relatedness will be assessed with this short form of the patient version of the WAI and is 12 items (e.g., We agree on what is important for me to work on.). The item scores will be averaged and the scale is 1 (Never) to 7 (Always).
Change from baseline Recovery Assessment Scale (RAS) at 3 months | measured with clients at 3 months
  Recovery attitudes will be measured by the brief version of the Recovery Assessment Scale which is a 24 item measure with response options ranging from 1 (Strongly disagree) to 5 (Strongly agree).
Change from baseline Recovery Assessment Scale (RAS) at 6 months | measured with clients at 6 months
  Recovery attitudes will be measured by the brief version of the Recovery Assessment Scale which is a 24 item measure with response options ranging from 1 (Strongly disagree) to 5 (Strongly agree).
Change from baseline State Hope Scale | measured with clients at 3 months
  Hopefulness in recovery-oriented services will be evaluated using the State Hope Scale, which includes 12 items with response options ranging from 1 (Definitely false) to 4 (Definitely true).
Change from baseline State Hope Scale | measured with clients at 6 months
  Hopefulness in recovery-oriented services will be evaluated using the State Hope Scale, which includes 12 items with response options ranging from 1 (Definitely false) to 4 (Definitely true).
Change from baseline Person Centered Care (PCC) Subscale at 3 months | measured with clients at 3 months
  Perceived quality of care will be measured by Person Centered Care (PCC), one of the two sub-scales of the Quality of Mental Health Care Scale (client version) developed to assess how clients rate the quality of care they receive (e.g., Staff helped me take steps towards one of my personal goals) using a scale ranging from 0 (Never) to 5 (always).
Change from baseline Person Centered Care (PCC) Subscale at 3 months | measured with clients at 6 months
  Perceived quality of care will be measured by Person Centered Care (PCC), one of the two sub-scales of the Quality of Mental Health Care Scale (client version) developed to assess how clients rate the quality of care they receive (e.g., Staff helped me take steps towards one of my personal goals) using a scale ranging from 0 (Never) to 5 (always).
Change from baseline Strengths Model Social Determinants of Health Scale | measured with clients at 3 months
  Social determinants of health (SDOH) with different aspects of life will be measured with a scale developed by the Strengths Model Inc. as part of a Strength Assessment. The scale consists of 6 items measuring satisfaction with the client's housing, employment, education, supportive relationships, community involvement, and overall well-being using a scale ranging from 1 (Very dissatisfied) to 5 (Very satisfied).
Change from baseline Strengths Model Social Determinants of Health Scale | measured with clients at 6 months
  Social determinants of health (SDOH) with different aspects of life will be measured with a scale developed by the Strengths Model Inc. as part of a Strength Assessment. The scale consists of 6 items measuring satisfaction with the client's housing, employment, education, supportive relationships, community involvement, and overall well-being using a scale ranging from 1 (Very dissatisfied) to 5 (Very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Sadaaki Fukui, PhD, MSW, MA, Principal Investigator — Indiana University

IPD SHARING:
Plan to Share IPD: Yes
The National Institute of Mental Health (NIMH) Data Archive (NDA) will be used for subject level data sharing.
Supporting Information: Study Protocol, ICF
Time Frame: The research community will have access to data when the award ends or at the time of publication.
Access Criteria: Access to data in the NDA is controlled. Researchers seeking data from NDA are expected to meet data security measures and are asked to submit a Data Use Certification. All data access requests go through the NDA Data Access Committee. The standard NDA data access process allows access for one year and is renewable.
URL: https://nda.nih.gov/